CLINICAL TRIAL: NCT03423329
Title: Effect of Preoperative Oral Administration of Ibuprofen and Acetaminophen on the Anesthetic Efficacy of Buccal Infiltration During Vital Pulpotomy of Mandibular Primary Molars: A Prospective, Double-blinded, Randomized Controlled Trial
Brief Title: Effectiveness of Buccal Infiltration During Vital Pulpotomy After Administering Two Analgesic Premedications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Reham Abou El Fadl, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FDASU-REC R 071607
Record Dates: First submitted 2017-12-28; First posted 2018-02-06 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Intervention:Drug: Brufen & Placebo
  Brufen syrup 10 ml, once, 1 hour before local anesthesia
  Interventions: Drug: Brufen; Drug: Placebo for Brufen
- Group B (Experimental): Intervention: Drug: Cital and Placebo
  Cital Syrup 10 ml, once 1 hour before Local anesthesia
  Interventions: Drug: Cital; Drug: Placebo for Brufen
- Group C (Placebo Comparator): Intervention: Drug: Placebo
  Other names:
  (Placebo for Brufen) (Placebo for Cital)
  Sansovit Iron Multivitamin syrup, an orange-coloured, orange-flavoured
  Interventions: Drug: Brufen; Drug: Cital; Drug: Placebo for Brufen

INTERVENTIONS:
Drug: Brufen — Brufen Syrup
  Other Names: Advil; Nurfen
  Arms: Group A; Group C
Drug: Cital — Cital Cyrup
  Other Names: Paramol
  Arms: Group B; Group C
Drug: Placebo for Brufen — Sansovit Syrup
  Other Names: Placebo for Cital

SUMMARY:
This Randomized study was designed to assess and compare the effect of two analgesic premedications (Ibuprofen BP 100 mg/5 ml and Paracetamol 200 mg/5ml.) on the anesthetic efficacy of buccal infiltration in vital pulpotomy of primary mandibular molars in children . A multivitamin with the same color as the twp tested medications will be administered to children in the control group. Parents of eligible children will be informed about the nature of the procedure, the purpose of the study, any possible discomfort or risks and a signed informed consent will be obtained from them prior to enrollment.

DETAILED DESCRIPTION:
A total of 60 healthy children will be recruited from the outpatient clinic of the Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Ain Shams University.

Inclusion Criteria include: age group 7-9 years Without systemic or mental disorders. Who could be categorized as cooperative according to Wright's classification for child behavior Ability of child to understand the use of pain scales; Having at least one lower second primary molar with deep caries indicated for pulpotomy; Absence of any periapical or furcation radiolucency on radiographs, Absence of any signs of internal or external resorption on radiographs, A vital coronal pulp on access opening.

. Patients who had taken analgesics within 12 hours before administration of the study drugs or those having active pain, pulpitis or abscess related to the designated mandibular molar will not be included.

To ensure randomization and allocation concealment, children will be randomly assigned to the three groups using computer-generated numbers.

One operator will do pulpotomy for all participants and to ensure blinding, another author ( will give the premedication to children.Pain during pulpotomy will be assessed using Wong Baker FACES pain assessment tool.

ELIGIBILITY:
Inclusion Criteria:

1. age group 7-9 years
2. Patients medically free.
3. Patients who can be categorized as cooperative or potentially cooperative according to Wright's classification for child behavior
4. Patients able to understand the use of pain scales;
5. Having at least one lower second primary molar with deep caries indicated for pulpotomy;
6. A vital coronal pulp on access opening of designated molar.

Exclusion Criteria:

1. Patients with allergic reactions, sensitivity, or contraindications to any tested drugs
2. Patients who had taken analgesics within 12 hours before administration of the study drugs
3. Patients having active pain, pulpitis or abscess related to the designated mandibular molar.
4. Children with special health care needs or any systemic problems
5. Presence of periapical or furcation radiolucency on radiographs in relation to designated molar
6. Presence of of any signs of internal or external resorption on radiographs in relation to designated molar

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Pain/discomfort felt during vital pulpotomy of mandibular second primary molars | 75 minutes after drug administration
  Using Wong Baker FACES pain assessment tool Children will be asked to rate any pain felt during coronal access

OTHER OUTCOMES:
Pain /discomfort in carious mandibular primary second molar | Just before drug administration
  Using Wong Baker FACES pain assessment tool Children will be asked to rate any pain felt in designated molar before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Reham Abou El Fadl, DDS, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Other, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within one month after study completion

DOCUMENTS (1):
  • Study Protocol (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03423329/Prot_000.pdf